CLINICAL TRIAL: NCT02240316
Title: An Observational Study of Patients With Malignant Lymphomas Treated With MabThera® SC in Everyday Clinical Practice
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28886
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Lymphoma, B-Cell, Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Follicular NHL Cohort
- DLBCL Cohort

SUMMARY:
This observational study aims to assess the therapeutic responsiveness of MabThera SC in patients with malignant lymphomas under everyday clinical practice conditions. Patients with previously untreated CD-20 positive follicular non-Hodgkin's lymphoma (NHL) or previously untreated CD-20 positive diffuse large B-cell lymphoma (DLBCL) who are planned for therapy with MabThera SC according to the assessment of the physician will be prospectively enrolled for observation. No study specific measures are required; treatment and documentation will be performed according to usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged >=18 years
* Previously untreated CD-20 positive follicular NHL
* Previously untreated CD-20 positive DLBCL
* Planned therapy with MabThera SC according to the assessment of the physician (before the start and independent from this study)
* Suitability for the therapy with MabThera SC

Exclusion Criteria:

All contraindications, interactions and incompatibilities for therapy with MabThera SC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CD-20 positive, diffuse large cell B-cell non-Hodgkin lymphoma (DLBCL) and CD-20 positive follicular non-Hodgkin lymphoma (NHL)
Sampling Method: Non-Probability Sample
Enrollment: 688 (Actual)
Dates: Start 2014-07-08 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in both indications (DLBCL and follicular NHL) who have reached a complete remission (CR), including unconfirmed complete remission (CRu) | Up to 2 years

SECONDARY OUTCOMES:
Total response rate | Up to 2.5 years
Two-year progression-free survival rate for patients with follicular lymphoma under maintenance therapy | 2 years
Safety profile: incidence, nature, severity, and outcomes of all adverse events and pregnancies (composite outcome measure) | Up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Universitätsklinikum Essen; Klinik für Hämatologie, Essen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).